CLINICAL TRIAL: NCT06429384
Title: Y-3 Injection in the Treatment of Acute Ischemic Stroke Phase II Clinical Trial -- Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Clinical Trial
Brief Title: Y-3 Injection in the Treatment of Acute Ischemic Stroke Phase II Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongjun Wang, Chief Physician, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-3-LC-02
Record Dates: First submitted 2024-04-03; First posted 2024-05-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Y-3 low dose group (20 mg/ time, qd), medium dose group (40 mg/ time qd), high dose group (60mg/ time, qd) and placebo control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In a double-blind design, the researchers, the researchers involved in the trial effect evaluation, the data managers, the statistical analysts, and the subjects and their relatives or guardians were blind to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Y-3 low-dose group (20 mg/dose, qd) (Experimental): Y-3 injection 20mg diluted with about 250 ml normal saline, intravenous infusion, qd, continuous medication for 10 days.
  Interventions: Drug: Y-3 Injection/Y-3 blank injection
- Y-3 medium dose group (40 mg/dose, qd) (Experimental): Y-3 injection 40mg diluted with about 250 ml normal saline, intravenous infusion, qd, continuous medication for 10 days.
  Interventions: Drug: Y-3 Injection/Y-3 blank injection
- Y-3 high-dose group (60 mg/dose, qd) (Experimental): Y-3 injection 60mg diluted with about 250 ml normal saline, intravenous infusion, qd, continuous medication for 10 days.
  Interventions: Drug: Y-3 Injection/Y-3 blank injection
- Blank control group (Placebo Comparator): Y-3 blank injection 10ml was diluted with about 250 ml normal saline, intravenous infusion, qd, and continuous medication for 10 days.
  Interventions: Drug: Y-3 Injection/Y-3 blank injection

INTERVENTIONS:
Drug: Y-3 Injection/Y-3 blank injection — The first dose should be completed as soon as possible after randomization; The time from the second dose to the first dose shall not be less than 12h, but not more than 24h+1h; The time interval of each subsequent administration is 24h±1h;

SUMMARY:
The objective of this clinical trial was to explore the efficacy and safety of Y-3 injection at different doses in patients with acute ischemic stroke within 48 hours of onset.

A multicenter, randomized, double-blind, parallel, placebo-controlled trial design was designed to include 240 participants.

Subjects press 1:1:1: 1 ratio of patients were randomly divided into Y-3 low-dose group (20 mg/ time, qd), medium-dose group (40 mg/ time, qd), high-dose group (60mg/ time, qd) and placebo control group, with 60 cases in each group. Random stratification factors include:

Time of onset (≤24 hours, > 24 hours). The patients were treated for 10 consecutive days (10 times) and followed up to 90 days after the first dose.

The trial was divided into three phases: screening/baseline, treatment, and follow-up.

Screening/baseline period: Subjects enter the screening/baseline period for screening examination after signing the informed consent.

Treatment period: Eligible subjects were randomly assigned at a ratio of 1:1:1:1 to receive Y-3 injection low-dose group, medium-dose group, high-dose group and placebo control drug for 10 consecutive days (10 times), during which relevant examinations required by the protocol were conducted and safety was assessed.

Follow-up period: Participants who finished treatment were followed up until 90 days after the first dose.

Stroke-related scale scores were performed at 10, 30, and 90 days after first use of the investigational drug The scores of Montgomery Depression Rating Scale (MSAS) and Hamilton Anxiety Scale (HAMA) were performed on the 10th and 90th days after the use of experimental drugs. Adverse events were recorded during treatment and follow-up to further assess safety

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel, placebo-controlled trial design was designed to include 240 participants, who were randomly assigned to Y-3 low-dose group (20 mg/ time, qd), medium-dose group (40 mg/ time, qd), high-dose group (60 mg/ time, qd) and placebo control group in a ratio of 1:1:1:1. Each group had 60 cases.

Random stratification factors included: onset time (≤24 hours, > 24 hours).The patients were treated for 10 consecutive days (10 times) and followed up to 90 days after the first dose.

The trial was divided into three phases:screening/baseline, treatment, and follow-up.

Screening/baseline period: Subjects enter the screening/baseline period for screening examination after signing the informed consent.Treatment period: Eligible subjects were randomly assigned at a ratio of 1:1:1:1 to receive Y-3 injection low-dose group, medium-dose group, high-dose group and placebo control drug for 10 consecutive days (10 times), during which relevant examinations required by the protocol were conducted and safety was assessed.Follow-up period: Participants who finished treatment were followed up until 90 days after the first dose.Stroke-related scale scores were performed on the 10th, 30th and 90th days after the first use of the experimental drug, and Montgomery Depression Rating Scale (MADRS) and Hamilton Anxiety Scale (HAMA) scores were performed on the 10th and 90th days after the first use of the experimental drug. Adverse events were recorded during treatment and follow-up to further assess safety.

ELIGIBILITY:
Inclusion Criteria:

-

Only those who meet all the following criteria can be included in the group:

1. Age ≥ 18 years old and<81 years old, regardless of gender;
2. After the onset of this disease, the National Institutes of Research Stroke Scale score was 6 ≤ NIHSS ≤ 20 points, and the sum of the 5th upper limb and 6th lower limb scores was ≥ 2 points. If patients receiving thrombolysis treatment were screened and evaluated based on the NIHSS score after thrombolysis;
3. Within 48 hours (including 48 hours) of onset;
4. Diagnosed as ischemic stroke according to the "Key Diagnostic Points for Various Major Cerebrovascular Diseases in China 2019", with good recovery after the first or last onset (mRS score ≤ 1 point before this onset);
5. Obtain informed consent from the patient or their legal representative voluntarily signed and approved by the ethics committee.

Exclusion Criteria:

-

Those who meet one of the following criteria during filtering cannot be included in the group:

1. Intracranial hemorrhagic diseases seen on cranial imaging: hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc; If it is only oozing blood, the researcher can determine whether it is suitable for enrollment;
2. Severe consciousness disorder: The item score of NIHSS's 1a consciousness level is greater than 1 point;
3. Transient ischemic attack (TIA);
4. After controlling the patient's blood pressure, the systolic blood pressure remains ≥ 220mmHg or the diastolic blood pressure remains ≥ 120mmHg;
5. Previously diagnosed patients with severe mental disorders and severe dementia;
6. Patients previously diagnosed with depression or anxiety disorder;
7. Patients undergoing antidepressant or anti anxiety treatment;
8. Diagnosed with severe active liver diseases, such as acute hepatitis, chronic active hepatitis, liver cirrhosis, etc; Or ALT or AST>2.0 × ULN;
9. Diagnosed with severe active kidney disease or renal insufficiency; Or serum creatinine>1.5 × ULN;
10. After the onset of the disease, drugs with brain cytoprotection in the instructions have been used, such as edaravone, concentrated solution of edaravone and dextranol for injection, nimodipine, ganglioside, CDPC, piracetam, oxiracetam, butylphenylpeptide, human urinary kallidinogenase (Urinary Kallidinogenase), cinepazide, rat nerve growth factor, cerebrolysin (cerebroprotein hydrolysate), calf serum deproteinized injection Calf blood deproteinized extract injection, etc;
11. After the onset of this disease, thrombectomy or interventional therapy has been applied or planned to be applied;
12. Previously diagnosed with concurrent malignant tumors and undergoing anti-tumor treatment;
13. Previously diagnosed with severe systemic diseases, with an estimated survival period of<90 days;
14. The patient is in pregnancy, lactation, and there is a possibility of pregnancy in the patient/patient partner who plans to conceive during the trial period;
15. Previously known allergies to this product or any of its excipients (15-hydroxystearic acid polyethylene glycol ester, propylene glycol, sodium hydroxide);
16. A history of major surgeries within 4 weeks prior to enrollment and assessed by the researcher as affecting neurological function scores or affecting 90 day survival;
17. Have participated in other clinical studies or are currently participating in other clinical studies within the first 30 days of randomization;
18. The researcher believes that it is not suitable to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-06-04 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with mRS score ≤ 1 on the 90th day of treatment . | 90th day of treatment
  The proportion of subjects with mRS score ≤ 1 on the 90th day of treatment .

SECONDARY OUTCOMES:
Grade analysis of mRS Score on the 90th day of treatment; | 90th day of treatment
  Grade analysis of mRS Score on the 90th day of treatment;
The proportion of subjects with mRS Score ≤2 on the 90th day of treatment; | 90th day of treatment
  The proportion of subjects with mRS Score ≤2 on the 90th day of treatment;
Changes in NIH Stroke Scale from baseline on day 10 of treatment; | 10th day of treatment
  Changes in NIH Stroke Scale from baseline on day 10 of treatment;
Proportion of NIH Stroke of 0-1 or ≥4 reduction from baseline on day 10 and day 30 of treatment. | On the 10th and 30th day of treatment
  Proportion of NIH Stroke of 0-1 or ≥4 reduction from baseline on day 10 and day 30 of treatment.The content of NIHSS score included: consciousness level (consciousness level, consciousness level questioning, consciousness level command), gaze, visual field, facial paralysis, upper limb movement, lower limb movement, body aid movement, sensation, language, dysarthria, neglect. The score ranges from 0 to 42, with higher scores indicating more severe nerve damage.Score 0 to 1: normal or nearly normal Scores 1-4: mild stroke/minor stroke .5 to 15 points: moderate stroke .15-20 points: moderate to severe stroke Scores 21-42: severe stroke

OTHER OUTCOMES:
Montgomery Depression Rating Scale scores on day 10 and day 90 were &lt, respectively; Proportion of patients with scores of 12, ≥12, and ≥22; | On the 10th and 90th day of treatment
  Montgomery Depression Rating Scale scores on day 10 and day 90 were &lt, respectively; Proportion of patients with scores of 12, ≥12, and ≥22.There are 10 items in the scale, with a total score of 60 points. The higher the score, the higher the degree of depression. MADRS < 12 indicates no depressive symptoms, 12≤MADRS < 22 indicates mild depression, 22≤MADRS < 30 indicates moderate depression, and MADRS≥30 indicates severe depression.
Hamilton Anxiety Scale scores on day 10 and day 90 were &lt, respectively; Proportion of patients with scores of 7, ≥7, and ≥14. | On the 10th and 90th day of treatment
  Hamilton Anxiety Scale (HAMA) scores on day 10 and day 90 were &lt, respectively; Proportion of patients with scores of 7, ≥7, and ≥14.The scale used a 5-level scoring method, and the criteria for each level were: 0-asymptomatic; 1- Light; 2- Medium; 3- heavy; 4- Extremely heavy. The total score of Hamilton anxiety Scale is a very important basis to reflect the severity of patients' anxiety, that is, the less severe the disease, the lower the total score; The more severe the condition, the higher the total score. A total score of less than 7 is considered to have no symptoms of anxiety; A score of 7-13 is considered to be likely to have anxiety; A score of 14 to 20 is considered to be definitely anxious; 21 to 28 points, is considered to have significant anxiety; A score greater than 29 is considered likely to be severe anxiety.
Incidence of adverse events (AE) in each group; | From the time the subject receives medication to the end of the 90th day of the treatment
  Incidence of adverse events (AE) in each group;
The incidence of treatment-related adverse events (TEAEs) in each group; | From the time the subject receives medication to the end of the 90th day of the treatment
  The incidence of treatment-related adverse events (TEAEs) in each group;
The occurrence of important adverse events in each group; | From the time the subject receives medication to the end of the 90th day of the treatment
  The occurrence of important adverse events in each group;
The occurrence of serious adverse events (SAEs) in each group; | From the time the subject receives medication to the end of the 90th day of the treatment
  The occurrence of serious adverse events (SAEs) in each group;
The occurrence of suspicious and unexpected serious adverse reactions (SUSAR) in each group; | From the time the subject receives medication to the end of the 90th day of the treatment
  The occurrence of suspicious and unexpected serious adverse reactions (SUSAR) in each group;
Laboratory examination indicators: blood routine, urine routine, blood biochemistry, Laboratory examination indicators: blood routine, urine routine, blood biochemistry, coagulation function | Baseline period, on the 10th , 30th and 90th day
  Detect blood routine through a blood cell analyzer, including white blood cell count, neutrophil count, lymphocyte count, hemoglobin, and platelet count.Use a biochemical analyzer to detect blood biochemistry, including alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, direct bilirubin, creatinine, urea/urea nitrogen, uric acid, and so on. Detect coagulation function through a coagulation analyzer, including prothrombin time (PT), partially activated prothrombin time (APTT), international standardized ratio (INR), fibrinogen (FIB).Detect urine routine through a urine analyzer.These indicators are measured during the baseline period and post administration visit period to observe the impact of the drug on this indicator, whether the drug will cause AE and SAE，the occurrence of AE and SAE, the type and severity of AE and SAE, and ultimately to determine the safety of the drug.
Vital signs: heart rate, blood pressure, body temperature, respiration | Baseline period, on the 10th , 30th and 90th day
  Detecting parameters such as heart rate, electrocardiogram, and QT interval through an electrocardiogram monitor.Detecting blood pressure through a blood pressure monitor.Detecting body temperature through a thermometer.Detect respiratory rate by observing changes in chest contour count of the subject.These indicators are measured during the baseline period and post administration visit period to observe the impact of the drug on this indicator, whether the drug will cause AE and SAE，the occurrence of AE and SAE, the type and severity of AE and SAE, and ultimately to determine the safety of the drug.
Physical examination of the whole body: lungs, gastrointestinal tract, urinary system, musculoskeletal system, skin, lymph nodes, and other systems. | Baseline period, on the 10th , 30th and 90th day
  Detect systems such as lungs, gastrointestinal tract, urinary system, musculoskeletal, skin, lymph nodes, etc. through observation, auscultation, percussion, palpation, and other examination methods. These indicators are measured during the baseline period and post administration visit period to observe the impact of the drug on this indicator, whether the drug will cause AE and SAE，the occurrence of AE and SAE, the type and severity of AE and SAE, and ultimately to determine the safety of the drug.
Clinical laboratory examination | From the baseline period to the end of the 90th day of the treatment
  Laboratory evaluation not specified in the protocol, including parameters such as hematology, biochemical tests, urine analysis, etc. These indicators are measured during the baseline period and post administration visit period to observe the impact of the drug on this indicator, whether the drug will cause AE and SAE，the occurrence of AE and SAE, the type and severity of AE and SAE, and ultimately to determine the safety of the drug.
Discontinuation due to adverse events; | From the beginning to the end caused by adverse events
  Discontinuation due to adverse events【AE includes abnormal laboratory test results (haematological, clinical biochemical, or urinalysis) or other safety assessments (e.g. electrocardiograms, radiological scans, vital signs measurements), including deterioration relative to baseline and deemed clinically significant in the medical and scientific judgment of the investigator; Exacerbation of pre-existing diseases; A new condition detected or diagnosed after the initiation of the investigational drug.】
Discontinuation due to any other non-adverse event. | From the beginning to the end due to unexpected circumstances except for adverse events
  Discontinuation due to any other non-adverse event(Any discontinuation other than an adverse event)

CONTACTS AND LOCATIONS:
Overall Officials: Shuya Li, Study Director — IRB of Beijing Tiantan Hospital Capital Medical University Beijing
Locations (30):
- China (30):
  - Beijing Tiantan Hospital, Capital Medical University Beijing, Beijing, Beijing Municipality
  - Liuzhou Workers Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Nanyang Second People's Hospital, Nanyang, Henan
  - Nanyang South Stone Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Inner Mongolia Baotou Steel Hospital, Baotou, Inner Mongolia
  - Inner Mongolia International Mongolian Medicine Hospital, Hohhot, Inner Mongolia
  - Huai 'an First People's Hospital, Huai'an, Jiangsu
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Lianyungang Second People's Hospital, Lianyungang, Jiangsu
  - Taizhou Second People's Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital (Old Hospital Area), Xuzhou, Jiangsu
  - Xuzhou Central Hospital（New compound）, Xuzhou, Jiangsu
  - Xuzhou First People's Hospital, Xuzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Beipiao Central Hospital, Beipiao, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Chinese People's Liberation Army Northern Theater Command General Hospital, Shenyang, Liaoning
  - Shenyang First People's Hospital, Shenyang, Liaoning
  - Shandong Third Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Tancheng County First People's Hospital, Linyi, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Dongyang City People's Hospital, Dongyang, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Result] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Result] van Horn N, Kniep H, Leischner H, McDonough R, Deb-Chatterji M, Broocks G, Thomalla G, Brekenfeld C, Fiehler J, Hanning U, Flottmann F. Predictors of poor clinical outcome despite complete reperfusion in acute ischemic stroke patients. J Neurointerv Surg. 2021 Jan;13(1):14-18. doi: 10.1136/neurintsurg-2020-015889. Epub 2020 May 15. PMID 32414889
- [Result] Lee SH, Kim BJ, Han MK, Park TH, Lee KB, Lee BC, Yu KH, Oh MS, Cha JK, Kim DH, Nah HW, Lee J, Lee SJ, Kim JG, Park JM, Kang K, Cho YJ, Hong KS, Park HK, Choi JC, Kim JT, Choi K, Kim DE, Ryu WS, Kim WJ, Shin DI, Yeo M, Sohn SI, Hong JH, Lee J, Lee JS, Khatri P, Bae HJ. Futile reperfusion and predicted therapeutic benefits after successful endovascular treatment according to initial stroke severity. BMC Neurol. 2019 Jan 15;19(1):11. doi: 10.1186/s12883-019-1237-2. PMID 30646858
- [Result] Meyer L, Alexandrou M, Leischner H, Flottmann F, Deb-Chatterji M, Abdullayev N, Maus V, Politi M, Roth C, Kastrup A, Thomalla G, Mpotsaris A, Fiehler J, Papanagiotou P. Mechanical thrombectomy in nonagenarians with acute ischemic stroke. J Neurointerv Surg. 2019 Nov;11(11):1091-1094. doi: 10.1136/neurintsurg-2019-014785. Epub 2019 Apr 27. PMID 31030188
- [Result] Chamorro A, Lo EH, Renu A, van Leyen K, Lyden PD. The future of neuroprotection in stroke. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):129-135. doi: 10.1136/jnnp-2020-324283. Epub 2020 Nov 4. PMID 33148815
- [Result] Li J, Zhang L, Xu C, Shen YY, Lin YH, Zhang Y, Wu HY, Chang L, Zhang YD, Chen R, Zhang ZP, Luo CX, Li F, Zhu DY. A pain killer without analgesic tolerance designed by co-targeting PSD-95-nNOS interaction and alpha2-containning GABAARs. Theranostics. 2021 Apr 3;11(12):5970-5985. doi: 10.7150/thno.58364. eCollection 2021. PMID 33897893
- [Result] Li J, Zhang L, Xu C, Lin YH, Zhang Y, Wu HY, Chang L, Zhang YD, Luo CX, Li F, Zhu DY. Prolonged Use of NMDAR Antagonist Develops Analgesic Tolerance in Neuropathic Pain via Nitric Oxide Reduction-Induced GABAergic Disinhibition. Neurotherapeutics. 2020 Jul;17(3):1016-1030. doi: 10.1007/s13311-020-00883-w. PMID 32632774
- [Result] Kaur H, Prakash A, Medhi B. Drug therapy in stroke: from preclinical to clinical studies. Pharmacology. 2013;92(5-6):324-34. doi: 10.1159/000356320. Epub 2013 Dec 12. PMID 24356194
- [Result] Fisher M; Stroke Therapy Academic Industry Roundtable. Recommendations for advancing development of acute stroke therapies: Stroke Therapy Academic Industry Roundtable 3. Stroke. 2003 Jun;34(6):1539-46. doi: 10.1161/01.STR.0000072983.64326.53. Epub 2003 May 15. PMID 12750546
- [Result] Hackett ML, Kohler S, O'Brien JT, Mead GE. Neuropsychiatric outcomes of stroke. Lancet Neurol. 2014 May;13(5):525-34. doi: 10.1016/S1474-4422(14)70016-X. Epub 2014 Mar 28. PMID 24685278
- [Result] Ferro JM, Caeiro L, Figueira ML. Neuropsychiatric sequelae of stroke. Nat Rev Neurol. 2016 May;12(5):269-80. doi: 10.1038/nrneurol.2016.46. Epub 2016 Apr 11. PMID 27063107
- [Result] Murrough JW, Abdallah CG, Mathew SJ. Targeting glutamate signalling in depression: progress and prospects. Nat Rev Drug Discov. 2017 Jul;16(7):472-486. doi: 10.1038/nrd.2017.16. Epub 2017 Mar 17. PMID 28303025
- [Result] Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011 Apr;16(4):383-406. doi: 10.1038/mp.2010.120. Epub 2010 Nov 16. PMID 21079608
- [Result] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Result] Griebel G, Holmes A. 50 years of hurdles and hope in anxiolytic drug discovery. Nat Rev Drug Discov. 2013 Sep;12(9):667-87. doi: 10.1038/nrd4075. PMID 23989795
- [Result] Shabel SJ, Proulx CD, Piriz J, Malinow R. Mood regulation. GABA/glutamate co-release controls habenula output and is modified by antidepressant treatment. Science. 2014 Sep 19;345(6203):1494-8. doi: 10.1126/science.1250469. Epub 2014 Sep 18. PMID 25237099
- [Result] Li YF. A hypothesis of monoamine (5-HT) - Glutamate/GABA long neural circuit: Aiming for fast-onset antidepressant discovery. Pharmacol Ther. 2020 Apr;208:107494. doi: 10.1016/j.pharmthera.2020.107494. Epub 2020 Jan 25. PMID 31991195
- [Result] Gould TD, Zarate CA Jr, Thompson SM. Molecular Pharmacology and Neurobiology of Rapid-Acting Antidepressants. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:213-236. doi: 10.1146/annurev-pharmtox-010617-052811. Epub 2018 Oct 8. PMID 30296896
- [Result] Zhou L, Li F, Xu HB, Luo CX, Wu HY, Zhu MM, Lu W, Ji X, Zhou QG, Zhu DY. Treatment of cerebral ischemia by disrupting ischemia-induced interaction of nNOS with PSD-95. Nat Med. 2010 Dec;16(12):1439-43. doi: 10.1038/nm.2245. Epub 2010 Nov 21. PMID 21102461
- [Result] Luo CX, Lin YH, Qian XD, Tang Y, Zhou HH, Jin X, Ni HY, Zhang FY, Qin C, Li F, Zhang Y, Wu HY, Chang L, Zhu DY. Interaction of nNOS with PSD-95 negatively controls regenerative repair after stroke. J Neurosci. 2014 Oct 1;34(40):13535-48. doi: 10.1523/JNEUROSCI.1305-14.2014. PMID 25274829
- [Derived] Feng B, Li H, Xu S, Li J, Wang Y, Zhao X, Wei Y, Xiao X, Wang S, Wang Y, Li S. Loberamisal injection for the treatment of acute ischaemic stroke: a multicentre, randomised, double-blind, placebo-controlled phase II clinical trial. Stroke Vasc Neurol. 2025 Nov 10:svn-2025-004581. doi: 10.1136/svn-2025-004581. Online ahead of print. PMID 41218852